CLINICAL TRIAL: NCT05212701
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 2 Study to Assess Efficacy and Safety of Reparixin in Cancer Related Fatigue in Pts With Advanced / Metastatic Breast Cancer Undergoing Taxane-based Chemotherapy.
Brief Title: To Assess Efficacy and Safety of Oral Reparixin in Patients With Fatigue and Locally Advanced / Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Dompé decided to withdraw the study due to the numerous difficulties encountered in enrollment, mainly due to the rapidly and continuously changing oncology drug scenario . No patients were enrolled.
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REP0121; 2021-000382-32 (EudraCT Number)
Record Dates: First submitted 2021-12-29; First posted 2022-01-28 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Fatigue; Locally Advanced or Metastatic Breast Cancer
Keywords: metastatic breast cancer
MeSH Terms: conditions — Fatigue; Breast Neoplasms | interventions — reparixin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reparixin (Experimental): Reparixin will be administered orally at the dose of 1200 mg (2 x 600 mg tablets) three times daily (total dose of 3600 mg/day) with no interruptions during each cycle.
  Interventions: Drug: Reparixin
- Placebo (Placebo Comparator): Masked placebo will be administered orally (2 tablets) three times daily with no interruptions during each cycle.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Reparixin — The oral tablets of the investigational product (IP) will be administered with water prior to the start of the anticancer treatment infusion on Day 1 Cycle 1 and then administered approximately every eight hours (± 2 h) with a glass of water (about 250 mL) and a light meal or snack (it is preferable that reparixin is taken with food).
  Arms: Reparixin
Drug: Placebo — The oral tablets of masked placebo will be administered with water prior to the start of the anticancer treatment infusion on Day 1 Cycle 1 and then administered approximately every eight hours (± 2 h) with a glass of water (about 250 mL) and a light meal or snack
  Arms: Placebo

SUMMARY:
Primary objective:

• To assess the efficacy of reparixin compared to placebo in limiting CRF in adult patients with locally advanced or metastatic breast cancer undergoing single-agent taxane chemotherapy, using FACITFatigue scale.

The secondary objectives are:

* To evaluate change in Quality of Life in the two treatment arms
* To assess the percentage of patients treated with reparixin compared to placebo delaying and discontinuing chemotherapy
* To assess Patient Global Impression of Severity (PGI-S) score and Patient Global Impression of Change (PGI-C) score associated with reparixin compared to placebo
* To assess the effect of reparixin compared to placebo on ECOG PS
* To assess the effects of reparixin vs placebo on Objective Response Rate (ORR), Progression Free Survival (PFS), Overall Survival (OS)

The safety objective is:

• To assess the safety and tolerability of reparixin in adult patients undergoing taxane-containing chemotherapy.

The pharmacokinetic (PK) objective is:

• To define the PK profile of orally administered reparixin, its metabolites (DF2243Y, DF2188Y, ibuprofen) and concomitant antineoplastic agents (paclitaxel, or nab-paclitaxel or docetaxel) in adult patients with locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
This is a phase 2, multinational, multicenter, randomized, double-blind, placebo-controlled study. It will evenly randomize 68 evaluable men and women adult patients with CRF in locally advanced or metastatic breast cancer who are candidates to start single-agent taxane chemotherapy (paclitaxel, nab-paclitaxel or docetaxel). CRF will be assessed at baseline on a scale from 0 - 10 (with 10 being most severe), enrolling any patient who report a score of 1 - 6. Recruitment will be competitive among the study sites, until the planned number of patients is randomized. Patients will be assigned (1:1) to receive either oral reparixin treatment (1200 mg t.i.d. - treatment group) or masked placebo t.i.d. (control group). Randomization will be stratified by site and according to the type of chemotherapy (paclitaxel vs docetaxel vs nab-paclitaxel). Sparse blood samples will be collected in the whole population for reparixin (and metabolites), docetaxel, nab-paclitaxel, paclitaxel PK analysis. Reparixin or placebo will be administered for 16 weeks or until disease progression, withdrawal of consent or unacceptable toxicity, whichever occurs first. Following the completion of the treatment, or after premature discontinuation during the double-blind phase the patients will be followed up for safety assessments for an additional 30 days after last study therapy administration and will be followed for progressive disease and survival until twelve months after last enrolled subject off treatment, or until trial is terminated for other reasons, whatever occurs first.

Number of Patients Sixty-eight (68) evaluable adult patients with CRF with locally advanced or metastatic breast cancer who are candidates to receive single-agent taxane chemotherapy will be included in the study. Assuming that 10% of subjects will not be evaluable for primary analysis, a total of approximately 76 subjects is expected to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provide written informed consent before the initiation of any study-specific procedures
* 2. Male or female ≥18 years of age
* 3. Pathologically documented locally advanced (not amenable to surgical resection) or metastatic HER2-negative breast cancer
* 4. Candidate to receive cycle 1 of treatment with single-agent taxane-based chemotherapy (paclitaxel, nab-paclitaxel, docetaxel)
* 5. CRF score from 1 to 6 on a numeric rating scale (NRS) from 0 to 10, where 0 = no fatigue, 10 = worst possible fatigue, during the previous 24 hours and lasting for a minimum of 4 days
* 6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2
* 7. Life expectancy of at least 6 months as estimated by the investigator
* 8. Able to swallow and retain oral medication (intact tablet)
* 9. Adequate organ function (defined by the following parameters):

  1. Serum creatinine < 140 μmol/L (< 1.6 mg/dL) or creatinine clearance > 60 mL/min
  2. Serum hemoglobin ≥ 11 g/dL; absolute neutrophil count ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L.
  3. Serum bilirubin ≤ upper limit of normal (ULN), except patients with Gilbert's syndrome.
  4. Serum Alanine aminotransferase (ALT), aspartate transaminase (AST) ≤ 1.5 x ULN
  5. Alkaline phosphatase ≤ 2.5 x ULN
  6. prothrombin time (PT) or activated partial thromboplastin time (aPTT, PTT) ≤ULN
* 10. No known hepatitis B virus (not due to immunization), hepatitis C virus, human immunodeficiency virus-I and -II positive status
* 11. If a female of childbearing potential, have a negative serum β-human chorionic gonadotropin (β-hCG) serum pregnancy test and use a highly effective method to avoid pregnancy for the duration of the trial and for at least 6 months after completion of docetaxel, paclitaxel or nab-paclitaxel therapy. Males of reproductive potential should use effective contraception during treatment and for 6 months after the last dose of docetaxel, paclitaxel or nab-paclitaxel

Exclusion Criteria:

* 1. More than 1 prior systemic chemotherapy for advanced disease. Patients may have received hormone therapy and biological therapy (e.g. CDK4/6 inhibitors), either alone or in combination
* 2. Malabsorption syndrome or disease significantly affecting gastrointestinal function including but not limited to gastrectomy or gastric outlet obstruction
* 3. History or evidence of neurological or psychiatric disorder or any other concurrent medical condition or disease that, in the opinion of the investigator or Medical Monitor may influence understanding of study and informed consent procedures, would pose a risk to subject safety or would interfere with the study evaluation, procedures or completion
* 4. Positive severe acute respiratory syndrome coronavirus 2 (SARSCoV- 2) antigenic test performed through nasal swab
* 5. Treatment with any investigational agent within at least 28 days or 5 half-lives (whatever is shorter) prior to Visit 1, recovered from previous treatment toxicity to Grade1 or better
* 6. Brain metastases that are untreated or symptomatic, or require any radiation, surgery, or continued steroid therapy to control symptoms from brain metastases
* 7. Treatment with oral morphine greater than 60 mg a day or equivalent
* 8. Other causes of fatigue, including, but not restricted to:

  1. untreated hypothyroidism
  2. pituitary disorder
  3. insomnia
  4. alcohol abuse
  5. uncontrolled pain as defined by pain intensity greater than 3 on a NRS (0-10)
  6. chronic >G2 anemia
  7. uncontrolled cardiac disease or cardiovascular disorders
  8. acute infections
  9. major depressive disorder
  10. uncontrolled neurological disorders
* 9. Concomitant use of other medications/dietary supplements for fatigue
* 10. Concomitant use of cannabidiol (CBD) or Tetrahydrocannabinol (THC).
* 11. Any other invasive malignancy from which the patient has been disease-free for less than 5 years with the exception of curatively treated basal or squamous cell skin cancer
* 12. Patients who are committed to an institution by virtue of an order issued either by the judicial or the administrative authorities
* 13. Patients who are employees of the sponsor or investigator or otherwise dependent on them
* 14. History of:

  1. intolerance or hypersensitivity to paclitaxel, nab-paclitaxel, docetaxel or any other concomitant drug used in the study
  2. intolerance or hypersensitivity to ibuprofen or to non-steroidal anti-inflammatory drug (NSAIDs)
  3. intolerance or hypersensitivity to more than one medication belonging to the class of sulfonamides, such as sulfamethazine, sulfamethoxazole, sulfasalazine, nimesulide or celecoxib; hypersensitivity to sulphanilamide antibiotics alone (e.g. sulfamethoxazole) does not qualify for exclusion
  4. lactase deficiency, galactosaemia or glucose-galactose malabsorption
  5. documented allergic reaction or severe reaction of any kind to dairy products
* 15. Pregnancy or lactation or unwillingness to use adequate method of birth control. Effective contraceptive measures include intrauterine device (IUD), bilateral tubal occlusion, vasectomised partner, sexual abstinence.
* 16. Concomitant use of ibuprofen or CYP2C9 inhibitors/inducers and inability to pause these drugs during the study
* 17. Concurrent use of NSAIDs or inability to stop NSAIDs during the treatment period
* 18. Any contraindications to NSAIDs including but not limited to previous experience of asthma, urticaria, or allergic-type reactions after taking aspirin or other NSAIDs.
* 19. A history of gastrointestinal bleeding or perforation related to previous NSAIDs therapy or an active or history of recurrent peptic ulcer/haemorrhage, coagulation disturbances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in FACIT-F score | week 16
  The Functional Assessment of Chronic Illness Therapy - fatigue (FACIT-fatigue) scale is a 13-item instrument designed to assess fatigue/ tiredness and its impact on daily activities and functioning in a number of chronic diseases. The instrument includes items such as tiredness, weakness, listlessness, lack of energy, and the impact of these feelings on daily functioning (e.g., sleeping, and social activities).
  The FACIT-fatigue scale is a 13-item patient-reported measure of fatigue where items are scored on a 0 - 4 response scale with anchors ranging from "Not at all" to "Very much so". To score the FACIT-fatigue, all items are summed to create a single fatigue score with a range from 0 to 52, where higher scores represent better functioning or less fatigue.

SECONDARY OUTCOMES:
Change from baseline in FACIT-F score | weeks 4, 8 and 12
  The Functional Assessment of Chronic Illness Therapy - fatigue (FACIT-fatigue) scale is a 13-item instrument designed to assess fatigue/ tiredness and its impact on daily activities and functioning in a number of chronic diseases. The instrument includes items such as tiredness, weakness, listlessness, lack of energy, and the impact of these feelings on daily functioning (e.g., sleeping, and social activities).
  The FACIT-fatigue scale is a 13-item patient-reported measure of fatigue where items are scored on a 0 - 4 response scale with anchors ranging from "Not at all" to "Very much so". To score the FACIT-fatigue, all items are summed to create a single fatigue score with a range from 0 to 52, where higher scores represent better functioning or less fatigue.
EQ-5D-5L score | day 1 of each 21- or 28-day cycle, off treatment visit (or withdrawal), which means up to 70 weeks
  The EQ-5D-5L consists of 2 pages: the EQ-5D-5L descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box of the most appropriate statement in each of the 5 dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the 5 dimensions can be combined into a 5-digit number that describes the patient's health state.The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS is used as a quantitative measure of health outcome that reflect the patient's own judgment.
Patient Global Impression of Severity (PGI-S) score | day 1 of each 21- or 28-day cycle, off treatment visit (or withdrawal) which means up to 70 weeks
  The PGI-S is designed to capture subject's perception of overall symptom severity at the time of completion on a 5-point categorical response scale: "Please choose the response below that best describes the severity of your fatigue over the past week" and is scored from 1 to 5, with 1 indicating "None", 2 "Mild", 3 "Moderate", 4 "Severe", 5 "Very Severe". The higher the score, the worse the outcome.
Patient Global Impression of Change (PGI-C) score | day 1 of each 21- or 28-day cycle except for cycle 1, off treatment visit (or withdrawal), which means up to 70 weeks
  The PGI-C is designed to capture the subject's perception of change in their overall symptom severity from baseline until the time of completion. Change in severity is captured using a 5- point scale: "Please choose the response below that best describes the overall change in your fatigue since you started receiving the taxane-based chemotherapy" and is scored from 1 to 5, with 1 indicating "Much better", 2 "A little better", 3 "No change", 4 "A little worse", 5 "Much worse". The higher the score, the worse the outcome.
Proportion of patients delaying next administration of chemotherapy due to CRF | throughout the study, up to 70 weeks
  Proportion of patients delaying next dosing of chemotherapy due to chronic renal failure (CRF)
Proportion of patients discontinuing chemotherapy due to CRF | throughout the study, up to 70 weeks
  Proportion of patients discontinuing chemotherapy due to chronic renal failure (CRF)
Change in Eastern Cooperative Oncology Group Performance Status (ECOG PS) | baseline, day 1 of each 21- or 28-day chemotherapy cycle, off treatment visit (or withdrawal) which means up to 70 weeks
  ECOG PS is graded as follow:
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead The higher the score, the worse the outcome.
Overall Response Rate (ORR) | Through study treatment, up to 70 weeks
  ORR is defined as the proportion of patients with best overall response of CR or PR according to RECIST 1.1.
Progression Free Survival (PFS) | Up to 12 months post-treatment
  PFS is defined as the time from the date of randomization until the date of the first documented progression or death due to any cause. PFS will be assessed based on local investigator assessment per RECIST 1.1.
Overall Survival (OS) | Up to 12 months post-reparixin discontinuation
  OS is defined as the time from date of first administration of study treatment until date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Minnella, MD, Study Director — Dompé Farmaceutici S.p.A
Locations (20):
- United States (2):
  - Waverly Hematology, Cary, North Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee
- Germany (4):
  - Kliniken Essen-Mitte, Klinik für Senologie/ Interdisziplinäres Brustzentrum, Essen
  - Praxis für Interdisziplinäre Onkologie & Hämatologie, Freiburg im Breisgau
  - Mammazentrum Hamburg am Krankenhaus Jerusalem, Hamburg
  - Klinikum Ernst von Bergmann, Frauenklinik, Potsdam
- Italy (14):
  - IRCCS Oncologico Istituto Tumori Giovanni Paolo II, Bari
  - Azienda Ospedaliero Universitaria di Bologna - Policlinico S. Orsola-Malpighi, Bologna
  - ASST-Spedali Civili di Brescia, Brescia
  - E.O. Ospedali Galliera, Genova
  - Istituto Scientifico Romagnolo per lo Studio e La Cura dei Tumori SRL IRCCS, Meldola (FC)
  - IRCCS - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera di Perugia, Ospedale Santa Maria della Misericordia, Perugia
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - "Azienda Unità Sanitaria Locale della Romagna Ospedale Infermi di Rimini", Rimini
  - Istituti Fisioterapici Ospitalieri- IFO - Istituto Regina Elena, Roma
  - Fondazione Policlinico Universitario A. Gemelli, IRCCS, Roma
  - "Azienda Ospedaliero Universitaria Sant'Andrea ", Roma
  - Ospedale Giuseppe Mazzini di Teramo, Teramo
  - A.O. "Pia Fondazione Cardinale Panico", Tricase